CLINICAL TRIAL: NCT04629157
Title: The LAVA (Lateral Flow Antigen Validation and Applicability) Study for COVID-19
Acronym: LAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 290989
Record Dates: First submitted 2020-11-04; First posted 2020-11-16 (Actual); Results first posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-09

CONDITIONS: This is a Pilot Study Which Aims to Assess the Validity and Applicability of Lateral Flow Assays (LFAs) Which Can be Used as a Point of Care Test for COVID-19; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Paired testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All patients entering the study will undergo paired testing of a lateral flow device using an anterior nasal swab and an RT-PCR using a nose and throat swab.
  Interventions: Device: Innova Lateral Flow Device

INTERVENTIONS:
Device: Innova Lateral Flow Device — The Innova Lateral Flow Device will be used on anterior nasal swab specimens and RT-PCR will be performed on nose and throat swabs.

SUMMARY:
This is a pilot study which aims to assess the validity and applicability of lateral flow assays (LFAs) which can be used as a point of care test for COVID-19. The study will focus on children admitted to hospital or planned to have a procedure for which they require an anaesthetic. RT-PCR is the current gold standard test for COVID-19, but it usually takes approximately 24-48 hours for a test result to be returned which can slow the clinical care given to a patient and can potentially increase the risk of healthcare worker (HWC) exposure to COVID-19. LFAs are a point of care test which can identify children who have a high viral load of COVID-19 and are performed using a more acceptable method of swabbing for children, just inside the nostril. Using LFA potentially enables the identification of infectious children with COVID-19 to aid with immediate care of patients and limiting HWC and other patients' contact with the virus. This study aims to assess the test failure rate and identify reasons for this which can be addressed. It also aims to assess the discomfort of both tests for children, provide a comparison between the time to LCA and RT-PCR result and provide data for a trial to adequately power a prospective trial comparing RT-PCR and LFA.

DETAILED DESCRIPTION:
During the ongoing COVID-19 pandemic, testing of children for COVID-19 has become an area of substantial need and intense scrutiny. The current gold-standard method for SARS-CoV-2 detection is the real time reverse transcriptase polymerase chain reaction (RT-PCR), performed on a sample from the respiratory system. This diagnostic test identifies fragments of viral RNA which are specific to SARS-CoV-2 and amplifies them. It can detect even relatively low levels of RNA in people who have contracted the virus but have not yet developed a high viral load or symptoms. It can also detect RNA after the live virus has cleared, but fragments of the virus' RNA remain. This test has a high analytical sensitivity and specificity. However, obtaining an adequate specimen is more difficult in children as the test is uncomfortable and not always well tolerated. This means that the diagnostic sensitivity is approximately 80%(1). Nevertheless, RT-PCR currently remains the most accurate method of detection of SARS-CoV-2. However, logistical issues around RT-PCR mean that the availability and usability of the test is reduced. This is due to a combination of factors including testing site capacity, processing capacity and the time taken to process and report the results by centralised laboratories. The net result is that the high sensitivity and specificity of PCR is offset by the time lag for result reporting. In acute hospitals, these delays can lead to poor patient flow through clinical areas, overuse of personal-protective equipment (PPE) or late recognition of nosocomial transmission. Thus, rapid testing is of particular importance in identifying highly infective individuals, for example people who are about to undergo a high-risk aerosol generating procedure, enter a crowded emergency room, or in rapid investigation of localised outbreaks.

Alternative methods and modalities of testing have therefore been explored, in particular the use of anterior nasal swabs to detect the SARS-CoV-2. Salivary RT-PCR is also under investigation(2, 3) but is affected by some of the limitations of performing RT-PCR on any sample, as described above. An alternative method of detection of SARS-CoV-2 is the use of antigen testing using a lateral flow assay (LFA)(4). Antigen-detection diagnostic test are designed to directly detect SARS-CoV-2 proteins produced by replicating virus in respiratory secretions. Most antigen rapid diagnostic tests use a sandwich immunodetection method using a simple-to-use lateral flow test format similar to a pregnancy test. Antigen detection tests have several advantages compared to RT-PCR; 1) it can be performed on an anterior nasal swabs- a specimen which is much more acceptably obtained in children-, 2) the results can be rapidly processed using a commercial kit at the bedside, with a result being available within 30 minutes of the sample being taken, and 3) it is less expensive to perform an antigen test compared to RT-PCR. The trade-off for ease-of-use and rapid turnaround time of antigen tests is a decrease in sensitivity compared to RT-PCR, particularly if the person has a low viral load (e.g. they are early or late in the disease) because the levels of antigens present in the upper respiratory tract might fall below the threshold for detection. The analytical sensitivity appears to be approximately 50% overall, but this increases during periods of anticipated infectivity when the viral load is >60,000 (RT-PCR cycle time threshold <27) to approximately 90%. The specificity of antigen tests has consistently been reported to be very high (>97%). Thus, if the antigen test is positive then it is very likely that it is a true result, and the person does have COVID-19. Antigen-detection tests are therefore primarily being used to detect infectivity of an individual, rather than being used as a clinical diagnostic test for COVID-19.

The potential application of LFAs to defeat Covid-19 are evident, with several clinical scenarios below demonstrating areas where comparing the performance of RT-PCR to LFA could improve the care of children and improve the safety of staff in hospital. However, evaluation of the use of these tests in clinical settings is essential before full implementation in routine clinical practice is advised.

At present, all children are tested for COVID-19 with RT-PCR when they are admitted to hospital, regardless of their symptoms. During the winter months, when more children with respiratory symptoms will seek medical care, current guidance recommends isolation or cohorting of these patients within hospital until their SARS-CoV-2 test is back(5). However, the majority of children are likely to have an alternative cause for their symptoms, such as respiratory syncytial virus, adenovirus or influenza. Early identification of infectious children with COVID-19 using a point of care test would allow for more effective cohorting or isolation to occur and potentially reduce the spread of COVID-19 in hospital settings, not just from children but their parents too who are likely to be infected as a household contact. Besides, early identification of children with COVID-19 using LFA will aid compliance with stringent use of PPE for healthcare workers caring for these children.

Children being admitted for elective procedures are currently also routinely tested for COVID-19 with a nasopharyngeal swab prior to admission. This is performed to reduce the chance of them harbouring SARS-CoV-2 at the time of having a high-risk aerosol generating procedure (AGP), where the risk of transmission of SARS-CoV-2 to staff is increased. Generally, these children are asymptomatic, as the presence of ILI symptoms often precludes an anaesthetic being performed. In this population, LFAs could be used to identify children who were incubating SARS-CoV-2 at the time of swabbing but were not shedding the virus who have subsequently progress to start shedding the virus (Table 1). Performing LFA potentially enables infectious children to be identified and can be used to guide decisions around proceeding with a procedure and the use of PPE in children when the procedure goes ahead.

Finally, LFAs could be used in 'high risk' hospital areas, particularly intensive care and high dependency units where high-risk AGPs are commonly performed and where children are more likely to have symptoms which are in-keeping with COVID-19. Surveillance of SARS-CoV-2 using RT-PCR is being performed routinely in some units, but a 24-48 hour delay in the result has minimal impact on practice around AGPs. LFAs may be utilised as a screening tool for infectious patients in these areas to support the use of appropriate PPE.

Further use of these tests could also be considered within health care worker (HCW) screening for infectivity after known exposures to Covid-19 cases, to limit the number of HCW absences due to potential exposure both outside and inside the hospital. They could potentially also be used in the community, in settings such as schools and sports clubs, to identify infectious individuals. Validation and usability in a controlled clinical setting is recommended prior to use in the wider community. Mathematical analysis of LFAs shows that, due to their high specificity, the negative predictive value is good in times of both high and low prevalence, even when the sensitivity of the test is low.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 0 - <18 years undergoing combined nose and throat swabbing for an elective diagnostic or surgical procedure.
2. Children aged 0 - <18 years undergoing combined nose and throat swabbing on admission to hospital when there is a differential diagnosis of COVID-19.
3. Children aged 0 - <18 years undergoing routine combined nose and throat swabbing during a stay on the intensive care unit, the high dependency unit or a transplant ward.

Exclusion Criteria:

None

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Alder Hey in the Park, Liverpool
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside of the research team

REFERENCES:
- [Derived] Harwood R, Rad L, Kelly C, Shelton C, Shepherd E, Roderick M, Whittaker E, Dyke S, Patel SV, Gent N, Kenny SE. Lateral flow test performance in children for SARS-CoV-2 using anterior nasal and buccal swabbing: sensitivity, specificity, negative and positive predictive values. Arch Dis Child. 2023 Feb;108(2):137-140. doi: 10.1136/archdischild-2022-324353. Epub 2022 Sep 9. PMID 36657801

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 322
Completed | 322
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 276
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 276
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135
  Male | 141
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 276

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Test
Description: A pain score (Wong-Baker) will be used to assess the pain of performing an anterior nasal swab and a nose and throat swab. This is a visual analog score accompanied by facial expressions from a scale of 0 to 10 where 0 is no pain and 10 is severe pain. The score is given by a child if they are old enough to do this, or by their parents if they are not, immediately after the swab has been performed.
Time Frame: Immediately after test on the day of test
Population: Children with a mean age of 7.7 years (std dev 5.2 years) were included.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 276
units on a scale
  Anterior nasal swab - parental report | 0 [0 to 2]
  Anterior nasal swab - child report | 0 [0 to 2]
  Nose and throat swab - parent report | 6 [4 to 8]
  Nose and throat swab - child report | 4 [2 to 8]

ADVERSE EVENTS:
Time Frame: Data were collected over 4 weeks
Description: No variation from the clinicaltrials.gov definition
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/276
Serious Adverse Events (participants affected / at risk) | 0/276
Other Adverse Events (participants affected / at risk) | 0/276

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04629157/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04629157/ICF_001.pdf